CLINICAL TRIAL: NCT03723486
Title: Changes in the Intestinal and Oral Microbiome of Morbidly Obese Patients Undergoing Gastric Bypass Surgery in Relation to Insulin Resistance and Metabolic Syndrome
Brief Title: Bariatric Surgery: Microbiome & Diabetes
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Johane Allard, Professor, Gastroenterologist, University Health Network, Toronto
Other Study IDs: 15-8784-AE; TB2-138775 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2017-11-13; First posted 2018-10-29 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Obesity
Keywords: Morbidly obese; Insulin resistance; Metabolic syndrome; Intestinal microbiome; Gastric bypass; Oral microbiome
MeSH Terms: conditions — Obesity; Insulin Resistance; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples, blood samples, dental and tongue plaque, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Roux-en-Y gastric bypass surgery (RYGB): Morbidly obese patients undergoing gastric bypass surgery

SUMMARY:
This study is a prospective cohort study, following 80 morbidly obese patients undergoing bariatric surgery, specifically Roux-en-Y gastric bypass (RYGB). The investigators are measuring intestinal microbiota (IM) and oral microbiota (OM) at the beginning before any treatment, at the time of surgery, which is after a very low calorie standard diet, and 1 and 6 months after surgery. The investigators assess whether changes in IM are related to changes in insulin resistance (IR), other features of the metabolic syndrome (MetS) and OM.

DETAILED DESCRIPTION:
Morbid obesity is associated with not only type 2 diabetes (T2D) of morbidly obese patients), but also cardiovascular complications, all of which remarkably improved and even resolved with bariatric surgery, of which the RYGB surgery has become the gold standard. Many studies have shown that within a few weeks post-RYGB there is dramatic improvement in IR and/or T2D independent of weight loss that ensues. These results led us to hypothesize that changes in intestinal microbiome (IM) composition and metagenome may be independently associated with improvement in metabolic parameters in humans undergoing RYGB.

Another aspect of RYGB that has not been studied is the potential changes in oral microbiome (OM) and salivary proteome (SP) and their relationship with weight loss and metabolic improvement. Understanding the OM and SP in morbidly obese patients before and after RYGB is important because shifts in the OM and SP may explain the susceptibility of these patients for oral infections like periodontal disease, which is more prevalent and severe in this population, particularly if T2D is present To our knowledge there are no longitudinal studies the relation between oral and intestinal microbiome before and after bariatric surgery. Furthermore, there are no studies looking at the effect of weight-reduction with the very low calorie diet (VLCD) Optifast regimen on IM, which the investigators plan to do. As IM may contribute to obesity and IR/T2D, the latter being the most dominant feature of the MetS. However, whether specific IM compositions are associated with improvement of obesity, IR/T2D and other features of the MetS is not clear; and the effects of RYGB on IM for treatment of these disorders in morbid obesity have not been well studied.

The investigators will conduct a prospective observational study of morbidly obese patients undergoing RYGB, in which the investigators will measure the intestinal microbiome before and after surgery along with insulin resistance and metabolic syndrome. Baseline measurements will be done before the pre-operative run-in with the very low calorie Optifast regimen (800 kcal/d) given before the laparoscopic RYGB (1 week/100 lbs body weight) to reduce the liver size for surgical access. Preoperatively, Optifast likely leads to changes in IM (never assessed) in addition to weight loss and improvement in MetS parameters. Aim: To track the changes in IM structure and function (metagenome) of morbidly obese patients undergoing laparoscopic RYGB through 3 stages - a) before vs. after pre-op Optifast weight reduction treatment 24; and post-op RYGB at b) 1 month; and at c) 6 months. The investigators will correlate the specific changes in IM through these stages, to improvement in IR and other features of the MetS. At the same time points the investigators will also measure the OM, salivary flow rate and SP, as well as oral inflammatory load.

ELIGIBILITY:
Inclusion Criteria:

* Morbidly obese patients (BMI > 40 kg/m2 or BMI >35-40 kg/m2 with other severe weight loss responsive comorbidities, undergoing laparoscopic RYGB surgery).

Exclusion Criteria:

* regular intake of non-steroidal anti-inflammatory drugs; prebiotics, probiotics or antibiotics or any experimental drug in the 3 months prior to study entry; type 1 diabetes, chronic gastrointestinal diseases, previous gastrointestinal surgery modifying the anatomy, smoking; pregnancy or breastfeeding; patients not tolerating Optifast; bariatric surgery other than RYGB patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese patients undergoing RYGB surgery.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2015-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in HOMA-IR | Change from Baseline HOMA-IR at 6 months post bariatric surgery
  HOMA-IR which represents insulin resistance and is calculated based on (glucose [mmol/L] x insulin [mU/L] / 22.5).

SECONDARY OUTCOMES:
Stool Sample: 16S sequencing | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Stool sample analysis
Stool Sample: qPCR | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Stool sample analysis
Stool Sample: Short Chain fatty acid | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Stool sample analysis
Stool Sample: Metagenome. | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Stool sample analysis
Appetite assessment | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Appetite questionnaire
Anthropometry:Height | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Anthropometric height
Anthropometry: weight | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Anthropometric weight
Anthropometry: Waist circumference | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Anthropometric measurements (measured in cm)
Anthropometry: Hip-circumference | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Anthropometric measurements (measured in cm)
Questionnaires: Food record | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  General questionnaire
Questionnaires: Activity Log | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  General questionnaire
Questionnaires: Environmental questionnaire | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  General questionnaire
Questionnaires: Dental questionnaire, | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  General questionnaire
Oral microbiome: Saliva | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Oral sample
Oral microbiome: Mouth rinse | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Oral sample
Oral microbiome: Oral Plaque | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Oral sample
Oral microbiome: Tongue plaque | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Oral sample
C peptide | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Blood work measurements (measured in pmol/L)
HbA1c | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Blood work measurements (measured in %)
Glucose | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Blood work measurement (measured mmol/L)
Fasting Insulin | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Blood work measurement (measured in pmol/L)
Plasma endotoxin | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Blood work measurement of lipopolysaccharide
Gut Hormone | 4 time points; pre-Optifast (baseline), post-Optifast (at the time of surgery), 1 and 6 months post surgery
  Blood work measurement

CONTACTS AND LOCATIONS:
Overall Officials: Johane P Allard, MD, FRCPC, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto General Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Background] Lewis MC, Phillips ML, Slavotinek JP, Kow L, Thompson CH, Toouli J. Change in liver size and fat content after treatment with Optifast very low calorie diet. Obes Surg. 2006 Jun;16(6):697-701. doi: 10.1381/096089206777346682. PMID 16756727
- [Background] Chaffee BW, Weston SJ. Association between chronic periodontal disease and obesity: a systematic review and meta-analysis. J Periodontol. 2010 Dec;81(12):1708-24. doi: 10.1902/jop.2010.100321. Epub 2010 Aug 19. PMID 20722533
- [Background] Madsbad S, Dirksen C, Holst JJ. Mechanisms of changes in glucose metabolism and bodyweight after bariatric surgery. Lancet Diabetes Endocrinol. 2014 Feb;2(2):152-64. doi: 10.1016/S2213-8587(13)70218-3. Epub 2014 Feb 3. PMID 24622719
- [Background] Graessler J, Qin Y, Zhong H, Zhang J, Licinio J, Wong ML, Xu A, Chavakis T, Bornstein AB, Ehrhart-Bornstein M, Lamounier-Zepter V, Lohmann T, Wolf T, Bornstein SR. Metagenomic sequencing of the human gut microbiome before and after bariatric surgery in obese patients with type 2 diabetes: correlation with inflammatory and metabolic parameters. Pharmacogenomics J. 2013 Dec;13(6):514-22. doi: 10.1038/tpj.2012.43. Epub 2012 Oct 2. PMID 23032991
- [Background] Qin J, Li Y, Cai Z, Li S, Zhu J, Zhang F, Liang S, Zhang W, Guan Y, Shen D, Peng Y, Zhang D, Jie Z, Wu W, Qin Y, Xue W, Li J, Han L, Lu D, Wu P, Dai Y, Sun X, Li Z, Tang A, Zhong S, Li X, Chen W, Xu R, Wang M, Feng Q, Gong M, Yu J, Zhang Y, Zhang M, Hansen T, Sanchez G, Raes J, Falony G, Okuda S, Almeida M, LeChatelier E, Renault P, Pons N, Batto JM, Zhang Z, Chen H, Yang R, Zheng W, Li S, Yang H, Wang J, Ehrlich SD, Nielsen R, Pedersen O, Kristiansen K, Wang J. A metagenome-wide association study of gut microbiota in type 2 diabetes. Nature. 2012 Oct 4;490(7418):55-60. doi: 10.1038/nature11450. Epub 2012 Sep 26. PMID 23023125
- [Background] Le Chatelier E, Nielsen T, Qin J, Prifti E, Hildebrand F, Falony G, Almeida M, Arumugam M, Batto JM, Kennedy S, Leonard P, Li J, Burgdorf K, Grarup N, Jorgensen T, Brandslund I, Nielsen HB, Juncker AS, Bertalan M, Levenez F, Pons N, Rasmussen S, Sunagawa S, Tap J, Tims S, Zoetendal EG, Brunak S, Clement K, Dore J, Kleerebezem M, Kristiansen K, Renault P, Sicheritz-Ponten T, de Vos WM, Zucker JD, Raes J, Hansen T; MetaHIT consortium; Bork P, Wang J, Ehrlich SD, Pedersen O. Richness of human gut microbiome correlates with metabolic markers. Nature. 2013 Aug 29;500(7464):541-6. doi: 10.1038/nature12506. PMID 23985870
- [Background] Arimatsu K, Yamada H, Miyazawa H, Minagawa T, Nakajima M, Ryder MI, Gotoh K, Motooka D, Nakamura S, Iida T, Yamazaki K. Oral pathobiont induces systemic inflammation and metabolic changes associated with alteration of gut microbiota. Sci Rep. 2014 May 6;4:4828. doi: 10.1038/srep04828. PMID 24797416